CLINICAL TRIAL: NCT07160699
Title: To Evaluate the Effectiveness of an Interprofessional, Collaborative Approach to the Treatment of Spasticity Comprising Botulinum Toxin & Non-pharmacological Post-injection Therapy. A Study Protocol of a Multi-Centred N-of-1 Series
Brief Title: Effectiveness of an Interprofessional Approach to the Treatment of Spasticity With Botulinum Toxin & Non-pharmacological Therapies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Bern (Other)
Responsible Party: Principal Investigator, Clare Maguire, PhD Clinical Lead Physiotherapy, Technical University of Bern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00282
Record Dates: First submitted 2025-01-19; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Spasticity
Keywords: spasticity; neurorehabilitation; botulinium toxin; non-pharmacological interventions; multi-disciplinary
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: After the injection with BoNT, individualised, goal-specific non-pharmacological therapies will be provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapy with Botulinum Neurotoxin and non-pharmacological therapies (Experimental): Every included patient receive BoNT and non-pharmacological therpies. The participants serve as their own controls.
  Interventions: Drug: Botulinum Neurotoxin Type A; Other: Non-pharmacological therapies

INTERVENTIONS:
Drug: Botulinum Neurotoxin Type A — The effectiveness of the combination of BoNT with treatment goal specific non-pharmacological interventions will be evaluated.
Other: Non-pharmacological therapies — Depending on the treatment goal different non-pharmacological therapies as a standard of care will be provided
  Other Names: physiotherapy; occupational therapy

SUMMARY:
Many people with neurological conditions will experience spasticity, a nonvolitional and uncontrollable tightening and/or spasm of muscles. This can impact the person's functioning and independence in everyday tasks and can contribute to contractures. Spasticity and contracture develop and affect each person differently. Treatment is provided by a multi-disciplinary team (MDT), working collaboratively to offer the best combination of medications (including botulinum neurotoxin (BoNT)) and non-pharmacological interventions. There are a wide range of therapy interventions available. Each person's treatment plan is uniquely tailored to them, their individual presentation, and their treatment goals. Evidencing the effectiveness of spasticity and contracture treatment has been difficult. The manifestation and treatment of spasticity is never the same between patients. The experience of the condition and the perceived and observable effectiveness of treatment are unique to the individual. Treatment is most effective when MDT's work together to combine the most appropriate medications and therapies in a treatment plan individualised to the person and their presentation. Understanding how expert teams formulate spasticity treatment and how effectively their expertise influences spasticity outcomes could help inform practice.

The purpose of this multicenter, case study series is to evaluate the effectiveness of two conceptually similar, specialised MDT approaches for the treatment of patients with spasticity in two cross-national neurorehabilitation facilities.

The goal of this study is to investigate the effectiveness of interprofessional treatments of non-drug interventions in combination with botulinum toxin injections in patients who suffer from spasticity.

The main goals of the study are to evaluate:

1. Describe and evaluate the types of botulinum toxin and therapy treatment choices expert MDTs make when treating people with spasticity.
2. Evaluate whether a MDT approach to the assessment and treatment of spasticity using BoNT and non-pharmacological interventions is effective at achieving patient goals.
3. Evaluate whether a MDT approach to the assessment and treatment of spasticity using BoNT and non-pharmacological interventions, improves impairment and activity/participation outcomes using commonly used clinical outcome measures.

There will be no comparison group. The N-of-1, ABC study design allows participants to serve as their own controls.

Participants will undergo assessements to describe their goals and severity of spasticity:

* Goal Attainment Scale light
* ArmA & SQoL-6D
* LegA
* Modified Ashworth Scale
* Modifies Tardieu Scale
* Muscle Strength according to MRC
* Pain Measurement (NRS, VAS or other)

DETAILED DESCRIPTION:
Cross-national, multicenter (CH and UK) single case experimental design (SCED), specifically N-of-1 series with an ABC Design (Baseline, Intervention, Follow-up). Patients with focal or multifocal spasticity who the MDT determine that BoNT and concomitant therapies are appropriate interventions based on their multidisciplinary evaluation. As this is a trial with defined pharmacological and non-pharmacological interventions that are an integral part of the individual treatment, all measurements and treatments are included to varying degrees in the standard of care/usual care in the rehabilitation centres. Participants will receive their botulinum toxin and therapy treatments as recommended by their clinical team. Both are a standard care in rehabilitation of spasticity. Included patients receive their BoNT injection and non-pharmacological interventions as indicated. All participating patients will be repeatedly measured at baseline phase A (pre- intervention), during intervention phase B and after completion of the intervention during phase C follow-up. The repeated measurements at baseline allow the participants to serve as their own controls. With this method, the treatment efficacy for individual patients can be estimated, rather than aggregate group effects and therefore the true heterogeneity and varying responses of individual patients is captured.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* male, female or other
* acute or chronic spasticity
* patients who have been assessed by the spasticity MDT and whose treatment plan includes Botulinum toxin and non-pharmacological therapies for focal or multi-focal spasticity and who have signed the general consent at entry.

Exclusion Criteria:

* <18 years
* Patients with spasticity, who will not receive BoNT
* Planned re-injection of BoNT before the end of the Phase C Follow-Up
* Previous BoNT injection within 3 months of baseline measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale: A multidisciplinary team (MDT) approach to the assessment and treatment of spasticity using BoNT and non-pharmacological interventions, improve individualised, patient-centred functional outcomes based on collaborative goal setting | From enrollment: Baseline 2 weeks (4 times), Intervention 12 weeks (12 times), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  The Goal Attainment Scale (GAS) is a tool to formulate and measure personalized rehabilitation goals on all ICF levels. In this model the following 5-point rating is used:
  * 2 much better than defined
  * 1 better than defined 0 SMART formulated goal is achieved
    * 1 baseline status unchanged
    * 2 worsening of baseline status

SECONDARY OUTCOMES:
Leg Activity Measure (LegA): The influence on MDT approach on active or passive care of the affected limb | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (6x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  LegA: It is a valid and reliable tool, which measures change in passive and active function of the lower limb due to spasticity related impairment and the impact of these on quality of life. It is a patient or carer-rated outcome measure with 33 items relating to clinically relevant goals from the patient or carer's point of view. It is a 5 point Likert scale with 0 = no difficulties/ not at all and 4 = not able to do/ extremly.
Spasticity-related quality of life (SQoL-6D): Influence of the MDT approach on Quality of Life (QoL) | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (6x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  Spasticity-related quality of life (SQoL-6D) provides an overall picture of spasticity-related health status following focal treatment of upper limb spasticity. As a valid, reliable and responsive measure of spasticity-related quality of life, the SQoL is designed to record those dimensions that relate to the chosen goal areas. There are six dimensions of the SQoL-6D:
  1. Reduction of pain and discomfort
  2. Control of spasms and other involuntary movements
  3. Maintaining the range of upper limb movements
  4. Passive function: ease of caring for the affected limb
  5. Active function - using the affected limb in activities
  6. Mobility/ balance. Each dimension is assessed using a five-level scale ranging from 0 to 4, whereas 0 = no difficulties and 4 = extremly hard/ not able to do
Arm Activity Measure (ArmA): The influence on MDT approach on active or passive care of the affected limb | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (6x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  ArmA: It is a valid and reliable tool, which measures changes in passive and active function in the upper limb due to spasticity related impairment. It is a patient or carer rated outcome measure with 20 items relating to clinically relevant goals from the patient or carer's point of view. It is a 5-point Likert scale with 0 = no difficulties and 4 = not able to do.
  LegA: It is a valid and reliable tool, which measures change in passive and active function of the lower limb due to spasticity related impairment and the impact of these on quality of life. It is a patient or carer-rated outcome measure with 33 items relating to clinically relevant goals from the patient or carer's point of view. It is a 5 point Likert scale with 0 = no difficulties and 4 = not able to do.
Modified Ashworth Scale (MAS): The influence of the MDT approach on spasticity | From enrollment: Baseline 2 weeks (2-4times), Intervention 12 weeks (weekly), Follow-up 6 (1x) and 12 weeks (1x) after completion of intervention
  MAS: The MAS measures the severity of spasticity and is a six-point ordinal scale (0 - no difficulty, 4 - unable to do task) with an additional point at +1 (slight increase in muscle tone). The MAS therefore provides a single score to represent spasticity. It has moderate reliability but is widely used in clinical practice due to ease of application.
Modified Tardieu Scale (mTS): The influence of the MDT approach on spasticity | From enrollment: Baseline 2 weeks (2-4times), Intervention 12 weeks (weekly), Follow-up 6 (1x) and 12 weeks (1x) after completion of intervention
  mTS: The mTS is a reliable measure which quantifies spasticity by assessing the muscle response to different stretch velocities (movements at fast and slow speed passive movement) and by determining the spasticity angle. Additionally, the quality of muscle reaction regarding resistance, clonus or contracture is noted. It is a 5-point ordinal scale with 0=no resistance and 4=clonus > 10sec.
The influence of the MDT approach on muscle strength | From enrollment: Baseline 2 weeks (2-4 times), Intervention 12 weeks (weekly), Follow-up 6 (1x) and 12 weeks (1x) after completion of intervention
  Muscle strength will be tested manually by the examiner following the Medical Research Council (MRC) as a valid tool. The scale is an ordinal scale and ranges from 0-5 whereas grade 0 to 3 has the highest reliability and with score 0 (no strength at all) to 5 (maximum strength).
Pain - Numeric Rating Scale (NRS): Influence of the MDT approach on pain | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (12x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  For conscious patients the Numeric Pain Rating Scale (NRS) will be used. This scale measures the subjective intensity of pain. It is an 11-point scale scored from 0-10, whereas 0 = no pain and 10 = the most intense pain imaginable. It is described having a good sensitivity.
Pain - Zürich Observation Pain Assessment (ZOPA): Influence of the MDT approach on pain | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (12x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  The Zürich Observation Pain Assessment (ZOPA) is used to external assessment of pain in people with cognitive and/ or conscious impairments in the field of neurosurgery and neurology. The instrument consists of a defined pool of items (behavioural characteristics) and is divided into four categories with a total of 13 subcategories. It provides information about the presence of pain and not about the perceived pain quality. The scale is assessed in various dimensions (e.g. facial expressions, posture, verbal expressions), with each dimension being rated on a five-point scale from 0 (no expression) to 4 (highest degree of pain).
Pain - Behavioural Pain Assessment Tool: Influence of the MDT approach on pain | From enrollment: Baseline 2 weeks (4x), Intervention 12 weeks (12x), Follow-up 6 (1x) and 12 (1x) weeks after completion of intervention
  The behavioural pain assessment tool for patients in minimal conscious state will be used for the included patients at the Royal Hospital for Neuro-disability. It is a structured framework for recording and monitoring behaviours that may denote experience of pain in patients with prolonged disorders of consciousness. 7 items will be observed by a health-professional and then scored from 0 to 2. Whereas 0 means normal behaviour and 2 means a strong sign which can indicate stronger pain.

CONTACTS AND LOCATIONS:
Overall Officials: Margret Hund-Georgiadis, PD Dr.med., Study Director — REHAB Basel, Rehaklinik für Neurorehabilitation und Paraplegiologie
Locations (2):
- REHAB Basel, Basel, Switzerland
- Royal Hospital for Neuro-disability, London, West Hill Putney, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication